CLINICAL TRIAL: NCT04088240
Title: Effects of Omega-3 Docosapentaenoic Acid on Lipids and Other Risk Factors for Cardiovascular Disease
Acronym: DPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Supplements Expired
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ann Skulas-Ray, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1907850505
Record Dates: First submitted 2019-09-05; First posted 2019-09-12 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Elevated Triglycerides; Cardiovascular Risk Factor
Keywords: omega-3
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DPA enriched n-3 (Experimental): 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
  Interventions: Dietary Supplement: DPA enriched n-3
- n-3 control (Active Comparator): 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
  Interventions: Dietary Supplement: n-3 control
- Placebo (Placebo Comparator): 4 g/d placebo control ("light" olive oil)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DPA enriched n-3 — 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
  Arms: DPA enriched n-3
Dietary Supplement: n-3 control — 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
  Arms: n-3 control
Dietary Supplement: Placebo — 4 g/d placebo control ("light" olive oil)
  Arms: Placebo

SUMMARY:
Elevated plasma triglycerides (TG) are due to an excess of TG-rich lipoproteins of several different types, most commonly of very-low-density lipoproteins (VLDL), but also intermediate-density lipoproteins (IDL, or VLDL remnants), chylomicrons, and/or chylomicron remnants. Epidemiologic evidence that a moderate elevation in TG is often associated with increased atherosclerotic cardiovascular disease (ASCVD) risk, and more recent evidence from Mendelian randomization studies has shown that elevated TG associated with genetic variants may be a causal factor for ASCVD and possibly for premature all-cause mortality.[1-6] Fasting plasma TG concentrations may be categorized as: normal (< 150 mg/dL ), borderline (150-199 mg/dL), high TG (HTG, 200-499 mg/dL), and very high TG (VHTG, ≥ 500 mg/dL).[7, 8] Risk of acute pancreatitis is increased in VHTG patients, especially those with TG ≥ 1000 mg/dL.[9] For VHTG, the primary goal of therapy is to reduce TG to < 500 mg/dL,[10] whereas there is no specific treatment goal for HTG nor prescription indication. However, the omega-3 fatty acids, EPA and DHA have well-established efficacy in reducing TG in the range of 150-500 when administered at doses of > or = 3 g/d EPA+DHA (reviewed in Skulas-Ray et al. in press). Importantly, administration of omega-3 fatty acids to people with TG in this range lead to a 25% reduction in major adverse cardiovascular endpoints in the recently completed "Reduction of Cardiovascular Events with EPA Intervention Trial" (REDUCE-IT).[11]

The results of REDUCE-IT provide compelling evidence for the use 3 g/d omega-3 fatty acid supplementation to reduce cardiovascular risk among patients with TG 150-500 mg/dL. The concentrated EPA supplement used in REDUCE-IT is just one of three long chain n-3 omega-3 fatty acids that influence lipids and lipoproteins and other aspects of cardiovascular risk.

Most research has focused on the evaluation of EPA and DHA, which are the two predominant n-3 FA in fish and in n-3 agents, but docosapentaenoic acid (DPA) is present in fish oil, as well, and accumulates in the blood at similar concentrations. The carbon length of the n-3 FA appears important for physiological effects. EPA has a carbon length of 20, DHA has a carbon length of 22, and DPA, the metabolic intermediate of EPA and DHA, is a 22-carbon n-3 FA. DPA may have significant potential for treating HTG and VHTG,[12, 13] but research on this fatty acid remains limited. In a 2-week open-label crossover comparison of 4 g/d of a DPA concentrate (containing unspecified amounts of free DPA and EPA) vs. 4 g/d EPA concentrate in people with HTG, plasma TG were reduced 33% by the DPA concentrate, which was significantly more than the 11% reduction with EPA.[13] Thus, a recent scientific advisory from the American Heart Association (Skulas-Ray et al, in press) concluded that more research is needed to elaborate the lipid and lipoprotein effects of DPA.

Additional biomarker research suggests DPA similarly can influence health outcomes that respond to EPA and DHA. For instance, decreased serum concentrations of DPA and DPA + DHA have been associated with increased risk of risk of acute coronary events[14] and myocardial infarction[15], respectively. Plasma DPA was also inversely associated with incident cardiovascular disease (CVD) in some ethnic groups.[16]

In conclusion evidence supports a potential role of DPA in improving health, but results from clinical supplementation studies are needed to clarify the effect of DPA supplementation on lipids and lipoproteins as well as other cardiovascular disease risk factors-relative to supplementation with EPA and DHA-to ascertain whether enrichment of omega-3 concentrates with DPA could offer health benefits above and beyond concentrates that only contain EPA and DHA.

DETAILED DESCRIPTION:
This is a cross-over, double-blind, randomized, placebo-controlled clinical study. Each treatment phase will span a continuous 6-week period. Prior to the first treatment phase, participants will be assigned to receive the DPA enriched n-3 supplement, conventional n-3 supplement, and identical placebo in random order. A computer program will be used to randomly assign participants to a treatment sequence. After each treatment phase, participants will have a 2-week washout period before beginning the next treatment phase.

Intervention protocol and study treatments:

Study capsules will be provided bi-weekly at the Food, Bioactives, & Health Lab on the University of Arizona campus or the Collaboratory. Participants may schedule pick-up times that are most suitable for their schedules. A staff member will be available to meet with participants at each bi-weekly pick-up.

The treatments are as follows:

* 4 g/d DPA enriched n-3 concentrate (~980 mg DPA, 380 mg EPA, 1720 mg DHA)
* 4 g/d n-3 control (~980 oleic acid, 380 mg EPA, 1720 mg DHA)
* 4 g/d placebo control ("light" olive oil)

For each 6-week treatment phase, participants will consume 4 g/day of the DPA-enriched concentrate, n-3 matched control, or placebo control. Participants will be required to avoid consuming any other food or supplements that contain n-3 FA during treatment phases. They will also be asked to maintain their current dietary intake (with the exception of excluding additional n-3 containing foods or supplements) and maintain their physical activity level and body weight over the course of the study.

Each supplementation period will be at least 6 weeks in length. However, treatment periods can be extended by 2 weeks (up to 8 weeks total) to accommodate scheduling challenges due to illness, travel, etc. For example, should a participant be unable to come in on two separate mornings for testing after 6 weeks of supplementation, they may continue the supplement and schedule testing for the following week.

Screening:

Potential participants will be interviewed by telephone to determine their initial eligibility. If they remain eligible after the telephone screening, they will be further screened at the Collaboratory, CATS, or the Food, Bioactives, & Health Lab. This screening visit will consist of: filling out forms (informed consent, medical history, personal information); measuring height and weight so body mass index (BMI) can be calculated; and measuring blood pressure (BP). If it is determined that they are still eligible following these measurements, a blood sample will be taken and a complete blood cell count, health panel including liver and kidney function, and a blood fat panel will be performed (approximately 15 mL of blood or ~1 tablespoon will be taken). If the initial blood draw is unsuccessful, it may need to be repeated, with permission of the participant. Females of child-bearing age will be given a urine pregnancy test. Study investigators will review all of the screening data. Participants meeting eligibility criteria will be scheduled for baseline data collection and supplementation will begin thereafter.

Baseline and endpoint visits (4 total):

Participants will undergo additional clinical assessments for one day at baseline (screening values will be used as the second measure) and two days for each of 3 endpoint visits (at the end of each 6-week treatment phase). The baseline visit will be scheduled within 2 weeks of the participant's screening visit. Participants will be required to fast overnight (12 hours with no food or drink except water) and abstain from alcohol for 48 hours prior to each testing day. To ensure participant eligibility, a brief assessment will be administered (see ScreeningForm_DPA). If a participant does not meet the requirements, their visit will be rescheduled. Testing will be conducted at CATS, the Collaboratory, or the Food, Bioactives, & Health Lab and the procedures are described in more detail below.

• Blood sampling: Prior to having their blood taken, participants will be asked not to consume any food or drink except water for 12 hours and to avoid alcohol for 48 hours. Participants also should not engage in vigorous physical activity for 12 hours prior to having their blood taken. Two blood samples will be taken at baseline and at the end of each treatment phase (for a total of 8 times after eligibility screening). On two separate days, a blood sample will be taken from the participant's arm after a 12-hour fast (no food or drink except water). If the initial blood draw is unsuccessful it may need to be repeated, with the participant's permission. Approximately 60 mL (4 tablespoons) of blood will be collected at baseline and at the end of each treatment phase, over two days separated by at least 24 hours. This will be collected as ~52 mL on one day and ~7.5 mL on the other day. Throughout the entire study, blood will be taken 8 times for a total amount of ~247 mL (~16.5 tablespoons), including the blood taken for screening tests prior to the start of the study (~15 mL or 1 tablespoon).

* At the end of each testing period, blood will be tested for the following: glucose, insulin, triglycerides, HDL-C, non-HDL-C, and concentrations of inflammatory markers. Red blood cell fatty acid concentrations will also be measured to assess compliance.
* On an additional day at the end of each testing period, participants will provide a blood sample (~7.5 mL) to repeat lipid measurements, which can vary day-to-day.

Blood samples will be stored and analyzed after all participants have completed the study. Study results will be available after study completion (which may take 2 years or longer).

* Saliva Collection: Saliva samples will be collected using the passive drool technique. Participants will use the collection aid to pool saliva into a specialized 2 mL cryovial.
* Urine Pregnancy Testing: Female participants of childbearing age will be asked to provide a urine sample for pregnancy testing at baseline and at the end of each treatment phase. If a participant becomes pregnant, she will not be able to continue participating in the study.
* Pulse Wave Analysis (PWA): On one of the testing days for the baseline visit and at the end of each supplementation period, participants will undergo testing to measure their blood pressure and pulse waveforms. This will be assessed using the SphygmoCor System (AtCor Medical, Sydney, Australia). SphygmoCor testing will be performed prior to the fasting blood sample and at a consistent time (± 1 hour) for all baseline and endpoint visits. The PWA measurement is very similar to a routine blood pressure measurement and will be used to assess central blood pressure and wave reflection characteristics (augmentation index). These will be derived from brachial pressure waveforms using a validated generalized transfer function. PWA measurements will be taken following JNC7 blood pressure guidelines in a quiet, temperature-controlled, dimly lit room following a 5-minute seated rest period. Participants will be asked to sit quietly with their feet flat on the floor for at least 5 minutes. A blood pressure cuff will then be placed on the upper arm. The cuff will inflate, then deflate for 5 seconds, and then partially re-inflate. Participants will be asked to remain quiet and still during this measurement. The procedure will be repeated twice, for a total of 3 measurements, with approximately 1 minute of rest between each measurement. The last 2 results will be averaged to increase accuracy.
* Pulse Wave Velocity (PWV): Following the PWA measurement, participants will undergo an assessment of aortic stiffness, by measuring their carotid-femoral pulse wave velocity (PWV). For this measurement, participants will be asked to lay flat on a hospital bed without a pillow. Carotid and femoral arterial pressure waveforms will be measured simultaneously via an applanation tonometry sensor manually held in place above the right common carotid artery and a blood pressure cuff placed on the right common femoral artery. PWV will be calculated by dividing the linear distance between the carotid and femoral sites by the transit time using SphygmoCor system software. This test will be performed three times with approximately 1 minute between measurements, and the last 2 results will be averaged to increase accuracy.
* Heart Rate Variability (HVR): Following the PWV measurement, participants will undergo an assessment of cardiovascular health, by measuring their heart rate variability (HRV). For this measurement, participants will be asked to lay flat on a hospital bed without a pillow. Participants will be connected to the SphygmoCor system by 3 ECG leads placed on the upper torso. HRV information will be collected using SphygmoCor system software. This test will be performed three times with approximately 1 minute between measurements, and the last 2 results will be averaged to increase accuracy.

Midpoint Visits:

Supplements will be provided every 3 weeks at a designated study site on the University of Arizona campus or at the Collaboratory. Participants may schedule pick up times that work best with their schedule. A study staff member will be available at each pick up visit to meet with participants to answer questions or discuss side effects.

It will take approximately 22-28 weeks for participants to complete this research study. The total time for study visits at the Collaboratory, CATS, or the Food, Bioactives, & Health Lab after initial screening, is approximately 8 hours. Times may vary and pre-menopausal females will require an additional 5 minutes for a urine pregnancy test at screening, baseline, and the end of each treatment period. The following is an estimate of the amount of time participants will spend in study activities:

Screening appointment:

* Forms, blood pressure, and blood draw: 45-60 minutes
* Pregnancy testing (pre-menopausal females only): 5 minutes

Baseline:

* Endpoint testing:

  * Blood draw: 15 minutes
  * Saliva collection: 5 minutes
  * PWA/PWV/HRV testing: 45 minutes
  * Pregnancy testing (pre-menopausal females only): 5 minutes
* Second day of testing: (NA; lipid measurements from screening appointment will be used)

End of treatment periods 1, 2, and 3:

* Endpoint testing:

  * Blood draw: 15 minutes
  * PWA/PWV/HRV testing: 45 minutes
  * Pregnancy testing (pre-menopausal females only): 5 minutes
* Second day of testing:

  * Blood draw: 15 minutes
  * Saliva collection: 5 minutes *Day 1 and 2 measurements may be switched to accommodate participant schedules
* Visits every 3 weeks to pick up new supplements and return unused capsules: 15 minutes/visit (~90 minutes total)
* Daily consumption logs (completed at home): ~15 minutes total

Total time commitment: ~8-9 hours (8 visits for testing and approximately 6 visits to pick-up supplements, as well as completing logs at home) over the course of 22-28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elevated fasting TG (150-500 mg/dL)
* BMI of 18-40 kg/m2
* Consistent dosage for any medication/supplements taken for elevated lipids, blood pressure, glucose, or inflammatory conditions
* Ability to abstain from alcohol for 48 hours prior to lab testing
* Low fish consumption (<2 servings/week)

Exclusion Criteria:

* Pregnant or lactating
* Use of blood thinning medications
* Adherence to a weight loss program
* Allergy to fish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 6-8 weeks
  Fasting blood work (triglycerides)

SECONDARY OUTCOMES:
Pulse Wave Velocity (PWV) | 6-8 weeks
  As measured by SphygmoCor device
Augmentation Index | 6-8 weeks
  augmentation index corrected for heart rate
Other lipids | 6-8 weeks
  Fasting blood work (HDL-C, total cholesterol, and LDL-C)
Glucose | 6-8 weeks
  Fasting glucose
Insulin | 6-8 weeks
  Fasting blood work (insulin)
Non-HDL-C | 6-8 weeks
  Fasting blood work (non-HDL-C)
Central blood pressure | 6-8 weeks
  systolic and diastolic blood pressures

OTHER OUTCOMES:
DPA-derived pro-resolving lipid mediators | 6 weeks
  Fasting blood work (lipid mediators)
Inflammatory markers | 6-8 weeks
  Fasting blood work (CRP, TNF-α)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No